CLINICAL TRIAL: NCT03132415
Title: Get Connected: Linking YMSM to Adequate Care Through a Multilevel, Tailored WebApp Intervention
Brief Title: Get Connected Efficacy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of North Carolina (Other); University of Michigan (Other); University of Minnesota (Other); Emory University (Other); Children's Hospital of Philadelphia (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U19HD089881 (SubProject 8780); 1U19HD089881 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: Prevention & Control; Internet; Adolescents; Young adults
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Get Connected (Experimental): Get Connected is a brief intervention focused on resolving ambivalence about HIV prevention behaviors, increasing self-efficacy for change, and enhancing motivation moving toward action.
  Interventions: Behavioral: Get Connected
- HIV Test Locator (Active Comparator): Participants randomized to the control condition will receive the Get Connected testing site locator. Given the availability of search engines to locate HIV/STI testing sites, the test locator condition may be considered usual care.
  Interventions: Behavioral: HIV Test Locator

INTERVENTIONS:
Behavioral: Get Connected — The investigators designed the intervention to help participants increase their HIV risk awareness, promote self-appraisal and increase motivation for engaging in prevention services, problem solving barriers to accessing care, and locating culturally-sensitive providers. Intervention content is customized based on participants' socio-demographic characteristics, HIV/STI testing history and testing motivations, and recent sexual behaviors.
  Arms: Get Connected
Behavioral: HIV Test Locator — The investigators will use a HIV/STI testing locator as the attention-control condition. The test locator provides a list of HIV testing sites in a city or zipcode.
  Arms: HIV Test Locator

SUMMARY:
Get Connected (GC) is an online brief intervention that employs individual and systems-level tailoring technology to reduce barriers to HIV prevention care (e.g., HIV/STI testing, PrEP) for YMSM. The deployment of GC through a mobile-friendly WebApp seeks to optimize online interventions' acceptability, accessibility, availability, long-term affordability among youth. The investigators will enroll self-reported HIV-negative or sero-status unaware, sexually active YMSM (ages 15-24) across three cities and randomize them into the GC intervention condition or to an attention-control condition. Assessments will be collected at 30 days and at 3, 6, 9 and 12 month follow-up.

DETAILED DESCRIPTION:
The number of HIV infections among men who have sex with men aged 15-24 (YMSM) has grown significantly in the past decade. For YMSM to successfully engage in HIV prevention and care services requires that they navigate a series of multilevel barriers operating at the individual (e.g., risk awareness, self-efficacy to get tested), systems (e.g., costs, medical mistrust, lack of culturally competent care), and structural (e.g., homelessness, costs, stigma) levels.

The investigators developed Get Connected (GC) as an online brief intervention that employs individual and systems-level tailoring technology to reduce barriers to linkage to competent prevention care (e.g., HIV/STI testing, PrEP) for YMSM (ages 15-24). After a formative phase comprised of assessing HIV testing sites' performance via a mystery shopping procedure, the investigators will test the efficacy of GC for increasing YMSM's successful engagement in locally appropriate HIV prevention and care using a two-arm randomized controlled trial.

The trial will compare the full GC intervention to the GC HIV test locator. Participants will be recruited from three cities (Houston, Philadelphia and Atlanta) characterized by high HIV incidence, and followed over 12 months. Assessments will be collected at 30 days and at 3, 6, 9 and 12 month follow-up.

Specific Aims include:

Aim 1: Examine the quality of HIV test counseling and PrEP-related referrals to YMSM within local HIV/STI testing sites in 3 cities (Houston, Philadelphia & Atlanta).

Aim 2: Test the efficacy of GC for increasing HIV-negative or HIV-unknown YMSM's successful uptake of HIV prevention services (e.g., routine HIV/STI testing) and PrEP awareness and willingness, as compared to the attention-control condition over a 12-month period.

Aim 3: Qualitatively assess sites' satisfaction with performance assessments and their improvements in service delivery when working with YMSM across the three regions.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male sex at birth and currently identifies as male
* Aged 15 to 24 years (inclusive) at time of screening
* Self-report as HIV-negative or sero-status unaware
* Speak and read English
* Not be on PrEP at time of enrollment
* Report having consensual anal sex with a male partner in the prior 6 months
* Reside in Philadelphia, Houston, or Atlanta
* Access to internet

Exclusion Criteria:

* Assigned female sex at birth
* Assigned male sex at birth but identifies as transgender or gender non-conforming
* Aged 14 years or younger or 25 years or older at time of screening
* HIV-positive
* Does not speak or read English
* Currently taking PrEP
* Did not have consensual anal sex with a male partner in the prior 6 months
* Does not reside in Philadelphia, Houston, or Atlanta
* Currently incarcerated
* Planning to move out of the region in next 12 months

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, MD, Study Chair — University of North Carolina; Jose A Bauermeister, PhD, Principal Investigator — University of Pennsylvania; Rob B Stephenson, PhD, Principal Investigator — University of Michigan; Patrick S Sullivan, PhD, Study Chair — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset. Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the dataset. The de-identified data from this project will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Background] Bauermeister JA, Pingel ES, Jadwin-Cakmak L, Harper GW, Horvath K, Weiss G, Dittus P. Acceptability and preliminary efficacy of a tailored online HIV/STI testing intervention for young men who have sex with men: the Get Connected! program. AIDS Behav. 2015 Oct;19(10):1860-74. doi: 10.1007/s10461-015-1009-y. PMID 25638038
- [Background] Bauermeister JA, Pingel ES, Jadwin-Cakmak L, Meanley S, Alapati D, Moore M, Lowther M, Wade R, Harper GW. The use of mystery shopping for quality assurance evaluations of HIV/STI testing sites offering services to young gay and bisexual men. AIDS Behav. 2015 Oct;19(10):1919-27. doi: 10.1007/s10461-015-1174-z. PMID 26303197
- [Background] Horvath KJ, Bauermeister JA. eHealth Literacy and Intervention Tailoring Impacts the Acceptability of a HIV/STI Testing Intervention and Sexual Decision Making Among Young Gay and Bisexual Men. AIDS Educ Prev. 2017 Feb;29(1):14-23. doi: 10.1521/aeap.2017.29.1.14. PMID 28195779
- [Background] Bauermeister JA, Golinkoff JM, Horvath KJ, Hightow-Weidman LB, Sullivan PS, Stephenson R. A Multilevel Tailored Web App-Based Intervention for Linking Young Men Who Have Sex With Men to Quality Care (Get Connected): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Aug 2;7(8):e10444. doi: 10.2196/10444. PMID 30072358
- [Result] Bauermeister JA, Golinkoff JM, Lin WY, Claude KF, Horvath KJ, Dowshen N, Schlupp A, Vickroy WJ, Desir K, Lopez AV, Castillo M, Tanney M, Wimbly TA, Leung K, Sullivan PS, Santiago DL, Hernandez R, Paul ME, Hightow-Weidman L, Lee S, Stephenson R. Testing the Testers: Are Young Men Who Have Sex With Men Receiving Adequate HIV Testing and Counseling Services? J Acquir Immune Defic Syndr. 2019 Dec 1;82 Suppl 2(2):S133-S141. doi: 10.1097/QAI.0000000000002173. PMID 31658201
- [Derived] Bauermeister JA, Horvath KJ, Lin WY, Golinkoff JM, Claude KF, Dowshen N, Castillo M, Sullivan PS, Paul M, Hightow-Weidman L, Stephenson R. Enhancing routine HIV and STI testing among young men who have sex with men: primary outcomes of the get connected clinical randomized trial (ATN 139). BMC Public Health. 2024 Apr 17;24(1):1072. doi: 10.1186/s12889-024-18522-w. PMID 38632603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Get Connected | HIV Test Locator
Started | 143 | 142
Completed | 143 | 142
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Get Connected | HIV Test Locator | Total
Number analyzed (Participants) | 143 | 142 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.17 (1.986) | 21.11 (2.189) | 21.14 (2.086)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 143 | 142 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 27 | 57
  Not Hispanic or Latino | 113 | 115 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 19 | 14 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 31 | 52
  White | 89 | 74 | 163
  More than one race | 10 | 19 | 29
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Reporting Changes in Their HIV Testing Behavior Using Self-report Questionnaires
Description: The investigators will estimate the proportion of participants who test at least twice for HIV over a 12-month period by intervention group.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Get Connected | HIV Test Locator
Number analyzed (Participants) | 143 | 142
Participants | 53 | 54

2. Secondary Outcome: Percent of Participants Reporting Changes in PrEP Uptake Using Self-report Questionnaires
Description: The investigators will test the proportion of the sample that begins PrEP during the 12-month follow-ups.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Get Connected | HIV Test Locator
Number analyzed (Participants) | 143 | 142
Participants | 38 | 36

3. Secondary Outcome: Percent of Participants Reporting Changes in Their STI Testing Behavior Using Self-report Questionnaires
Description: The investigators will estimate the proportion of participants who test for STIs at least once over the trial period.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Get Connected | HIV Test Locator
Number analyzed (Participants) | 143 | 142
Participants | 73 | 75

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the year of study participation.
Arm/Group | Get Connected | HIV Test Locator
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/142
Other Adverse Events (participants affected / at risk) | 0/143 | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT03132415/Prot_SAP_000.pdf